CLINICAL TRIAL: NCT07139873
Title: A Phase 3, Open-Label, Randomized, Multicenter Study to Evaluate Anti-tumor Efficacy of DZD8586 Versus Investigator's Choice in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Study of DZD8586 Versus Investigator's Choice in r/r CLL/SLL (TAI-SHAN6)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dizal (Jiangsu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dizal Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZ2024B0002
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; idelalisib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily dose of DZD8586 (Birelentinib) (Experimental)
  Interventions: Drug: DZD8586
- Investigator's choice (Active Comparator)
  Interventions: Drug: Bendamustine; Drug: Idelalisib; Drug: Rituximab

INTERVENTIONS:
Drug: DZD8586 — Orally, 50 mg, once daily until treatment discontinuation criterion is met.
  Other Names: Birelentinib
  Arms: Daily dose of DZD8586 (Birelentinib)
Drug: Bendamustine — Administered intravenously
  Arms: Investigator's choice
Drug: Idelalisib — Administered orally
  Arms: Investigator's choice
Drug: Rituximab — Administered intravenously
  Arms: Investigator's choice

SUMMARY:
This is a phase 3, open-label, randomized, multi-center study assessing the efficacy and safety of DZD8586 versus investigator's choice in participants with chronic lymphocytic leukemia/small lymphocytic lymphoma who have progressed following prior therapy.

Primary objective of this study is to assess the efficacy using progression free survival assessed by independent review committee as primary endpoint. Approximately 250 participants are estimated to be randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥ 18 years of age.
2. ECOG performance status 0-2.
3. Confirmed diagnosis of relapsed or refractory CLL/SLL with indication for treatment.
4. Adequate bone marrow reserve and organ system functions.
5. Participants willing to comply with contraceptive restrictions.

Exclusion Criteria:

1. Any unresolved > Grade 1 adverse event at the time of starting study treatment.
2. Known or suspected Richter transformation.
3. Known or suspected CNS involvement.
4. Previous or current therapy and comedications meet exclusion criteria.
5. Participants with major cardiovascular disease, active infection, malignancy or uncontrolled systemic disease.
6. Nausea and vomiting not controlled or chronic gastrointestinal diseases, unable to swallow the formulated product or previous bowel resection that would preclude adequate absorption.
7. Women who are breast feeding.
8. History of hypersensitivity to active or inactive excipients of DZD8586 or drugs with a similar chemical structure or class.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) assessed by Independent Review Committee (IRC) | Approximately 36 Months

SECONDARY OUTCOMES:
PFS assessed by investigator | Approximately 36 Months
Objective response rate (ORR) by IRC and investigator | Approximately 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Dizal (Jiangsu) Pharmaceutical Co., Ltd.
Locations (2):
- China (2):
  - First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjing, Jiangsu
  - National Clinical Research Center for Blood Diseases, Blood Disease Hospital & Institute of Hematology, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No